CLINICAL TRIAL: NCT05937165
Title: Acute Bioavailability of Berry Flavonoids and Impact on Inflammatory Biomarkers in Older Adults With Minor Depressive Symptoms: A Pilot Study
Brief Title: ABSORB (Amount of Blueberries So Older Adults Reap Benefits)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00069826
Record Dates: First submitted 2023-06-29; First posted 2023-07-10 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Depressive Symptoms; Aging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Dose Freeze-dried Blueberry Powder (Active Comparator): Consumption of 24 g of freeze dried blueberry powder for 3 consecutive days.
  Interventions: Other: Freeze-dried Blueberry Powder
- Higher Dose Freeze-dried Blueberry Powder (Experimental): Consumption of 48 g of freeze dried blueberry powder for 3 consecutive days.
  Interventions: Other: Freeze-dried Blueberry Powder

INTERVENTIONS:
Other: Freeze-dried Blueberry Powder — Three day consumption of two doses of freeze-dried blueberry powder

SUMMARY:
This randomized, cross-over, pilot study aims to compare preliminary impact of a standard dose of blueberry powder (24 g) vs a higher dose (48 g) on the bioavailability of flavonoids and inflammatory biomarkers in older adults with minor levels of depressive symptoms.

DETAILED DESCRIPTION:
Blueberries are a rich source of anti-oxidants and dietary fiber, and are recommended to consume as a part of a healthy diet. Regular consumption of blueberries as a source of dietary antioxidants may be an effective way to lower inflammation in older adults, who commonly have higher levels of inflammatory markers. However, older adults typically have a decreased efficiency of nutrient absorption and may need a higher dose of blueberries to absorb enough of the flavonoids needed to reap their benefits on inflammation. Thus, it is important for preliminary studies to pre-determine an appropriate dose of blueberry flavonoids specifically for older adults. This study aims to evaluated the preliminary impact of freeze-dried blueberry powder consumption on flavonoid bioavailability and inflammatory biomarkers in older adults. This will be an individual-level, unblinded, randomized, cross over pilot study in 5 older adults with minor levels of depressive symptoms. Eligible participants will collect a 24 hour urine sample, and then come in for the baseline assessments and provide a blood sample. Next they will be randomized to consume either the higher dose (48 g/day, equivalent ~ 2 cups of fresh blueberries) or the lower dose (24 g/day, equivalent ~1 cup of fresh blueberries) for 3 days. After 3 days they will begin collecting a 24 hour urine sample, and come in to repeat the baseline assessments and provide a blood sample. After a two week wash out period, participants will repeat the same baseline and follow-up assessments while consuming the other powder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 years and older
* Minor levels of depressive symptoms (center for epidemiological studies depression scale, ≥4 and <16 points)

Exclusion Criteria*:

* Unwilling to follow the study protocol
* Cognitive impairment (assessed via the telephone Montreal Cognitive Assessment) defined as individuals scoring <19)
* Self-reporting a history of major depression, bipolar, schizophrenia, or other psychotic or neurologic disorders
* Self-reporting of history gastro-intestinal diseases/conditions e.g., of bowel resection, inflammatory bowel disease/syndrome, Celiac disease
* Self-reporting immune disorders, e.g., rheumatoid arthritis, cancer, and other immunocompromising conditions
* Self-reporting history of type 1 or type 2 diabetes
* Self-reporting any history of substance or alcohol use disorder
* Allergy to blueberries
* Self-reporting use of anti-inflammatory (e.g., fish oil or non-steroidal anti-inflammatory drugs) or immune-suppressant drugs
* Are excessive tea or coffee consumers (e.g., >3 cups/day)
* Recent and consistent use of antibiotics
* Currently taking or advised during the intervention to take anti-depressants
* Current homicidal or suicidal ideation (assessed via the P4 Suicidality Screener

  * All deviations must be approved by the study sponsor

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Freeze-dried Blueberry Powder (Standard Dose Then Higher Dose): Consumption of 24 g of freeze dried blueberry powder for 3 consecutive days and then consumption of 48 g of freeze dried blueberry powder for 3 consecutive days, separated by a washout.
- Freeze-dried Blueberry Powder (Higher Dose Then Standard Dose): Consumption of 48 g of freeze dried blueberry powder for 3 consecutive days and then consumption of 24 g of freeze dried blueberry powder for 3 consecutive days, separated by a washout.
Period: Overall Study
Arm/Group | Freeze-dried Blueberry Powder (Standard Dose Then Higher Dose) | Freeze-dried Blueberry Powder (Higher Dose Then Standard Dose)
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Freeze-dried Blueberry Powder (Standard Dose Then Higher Dose) | Freeze-dried Blueberry Powder (Higher Dose Then Standard Dose) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (4) | 76 (5) | 73 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6
Depressive Symptom Severity [Mean (Standard Deviation); unit: points] — Center for Epidemiological Studies Depression Scale - Revised (CESD-R). Scores range from 0-60 with higher points indicating more severe symptoms of depression.
  points | 3.0 (2.0) | 4.3 (3.1) | 3.7 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Urinary Flavonoid Biomarkers
Description: Change in total flavonoid metabolites found in the urine. The values for the metabolites represent the relative abundance of each metabolite, rather than absolute quantification, with higher values reflecting higher levels of total flavonoid metabolites in the urine.
Time Frame: Baseline and Day 3 of intervention
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Standard Dose Freeze-dried Blueberry Powder | Higher Dose Freeze-dried Blueberry Powder
Number analyzed (Participants) | 5 | 5
Unitless | 398863 (274183) | 1045795 (661053)

2. Primary Outcome: Inflammatory Biomarker C-reactive Protein
Description: Change in serum C-reactive Protein
Time Frame: Baseline and Day 3 of intervention
Measure: Mean (Standard Deviation); unit: nanograms/mL
Arm/Group | Standard Dose Freeze-dried Blueberry Powder | Higher Dose Freeze-dried Blueberry Powder
Number analyzed (Participants) | 5 | 6
nanograms/mL | -100 (642) | -635 (1318)

3. Secondary Outcome: Inflammatory Biomarker Tumor Necrosis Factor Alpha
Description: Change in tumor necrosis factor alpha
Time Frame: Baseline and Day 3 of intervention
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Standard Dose Freeze-dried Blueberry Powder | Higher Dose Freeze-dried Blueberry Powder
Number analyzed (Participants) | 5 | 6
picograms/mL | -0.03 (0.11) | 0.06 (0.08)

4. Secondary Outcome: Inflammatory Biomarker Interleukin 6
Description: Change in interleukin 6
Time Frame: Baseline and Day 3 of intervention
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Standard Dose Freeze-dried Blueberry Powder | Higher Dose Freeze-dried Blueberry Powder
Number analyzed (Participants) | 5 | 6
picograms/mL | 0.28 (0.55) | -1.3 (3.0)

5. Secondary Outcome: Inflammatory Biomarker Interferon Gamma
Description: Change in serum interferon gamma
Time Frame: Baseline and Day 3 of intervention
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: From enrollment until end of study visits, ~ 4 weeks
Groups:
- Standard Dose of Freeze-dried Blueberry Powder: Consumption of 24 g of freeze dried blueberry powder for 3 consecutive days
- Higher Dose of Freeze-dried Blueberry Powder: Consumption of 48 g of freeze dried blueberry powder for 3 consecutive days
Arm/Group | Standard Dose of Freeze-dried Blueberry Powder | Higher Dose of Freeze-dried Blueberry Powder
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

LIMITATIONS AND CAVEATS:
This data is used as hypothesis generating, and is a very small sample size. Interpret the results with caution.

The data for interferon-gamma is delayed due to the assay kit being back-ordered. We hope to submit these results by January 2026.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT05937165/Prot_SAP_000.pdf